CLINICAL TRIAL: NCT05698550
Title: The Role of Erzhi Tiangui Formula in Expected Poor Ovarian Responders Undergoing In Vitro Fertilization-Embryo Transfer: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Role of Erzhi Tiangui Formula in Expected POR Women Undergoing IVF-ET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shandong University of Traditional Chinese Medicine (Other)
Collaborators: The 960th Hospital of the PLA Joint Logistics Support Force (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Maternity and Child Health Care of Zaozhuang (Unknown); Yantai Shan Hospital (Unknown); Maternal and Child Health Care Hospital of Shandong Province (Unknown); Hospital for Reproductive Medicine Affiliated to Shandong University (Unknown); Chongqing Medical Center for Women and Children (Other); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Jing-Yan Song, Clinical Professor, Shandong University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDUTCMEZTG1104
Record Dates: First submitted 2023-01-11; First posted 2023-01-26 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Infertility, Female
Keywords: Erzhi Tiangui Formula; Poor ovarian response; In Vitro Fertilization and Embryo Transfer (IVF-ET); Advanced maternal age
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EZTG group (Experimental)
  Interventions: Drug: Erzhi Tiangui Granule
- Control group (Placebo Comparator)
  Interventions: Drug: Erzhi Tiangui Placebo

INTERVENTIONS:
Drug: Erzhi Tiangui Granule — The Drug Manufacturing Unit of the Affiliated Hospital of Shandong University of Traditional Chinese Medicine produced the EZTG granule.The EZTG was packaged as 3 g/bag, batch number 01-FZ032-03. The daily dose is equivalent to 15g of Ligustrum lucidum (Nv Zhen Zi),15g of Lotus japonicus (Han Lian Cao),15g of the fruit of Chinese wolfberry(Gou Qi Zi),15g of Cuscuta chinensis(Tu Si Zi), 15g of Radix Rehmanniae Preparata(Shu Di Huang),12g of Angelica sinensis(Dang Gui),12g of Paeonia lactiflora(Bai Shao),12g of Ligusticum wallichii(Chuan Xiong),12g of Rhizoma cyperi(Xiang Fu),and 9g of Radix Glycyrrhizae (Zhi Gan Cao).The placebo granule,which was Preparata mainly composed of dextrin, was made in a similar color and shape to EZTG.Placebo granules were packaged as 3g/bag, with the same package of the EZTG, batch number 01-FZ032-03-1. The EZTG or placebo was orally administered after being dissolved in water, 3g each time, 2 times a day.
  Arms: EZTG group
Drug: Erzhi Tiangui Placebo — The placebo consisted mainly of yellow bean powder, starch, carbogen, molasses and could mimic the appearance, color and smell of Erzhi Tiangui granules, but without any active ingredients. Daily doses of placebo were delivered in the same packaging as Erzhi Tiangui granules.
  Arms: Control group

SUMMARY:
This randomized controlled trial aims to determine whether Erzhi Tiangui Formula can optimize the reproductive outcomes of elderly patients with expected poor ovarian response, and to provide a new approach to traditional Chinese medicine assisted in vitro fertilization and embryo transfer (IVF-ET).

DETAILED DESCRIPTION:
In recent years, traditional Chinese medicine (TCM) has been involved with all aspects of assisted reproductive technology (ART), but it remains a long way from being applied to in vitro fertilization and embryo transfer (IVF-ET). Moreover, there is a lack of high-quality clinical research conducted on a large scale. The Erzhi Tiangui formula, which originated from Gui-Cheng Xia, a national TCM master, was composed and established by Professor Fang Lian, who was a national famous TCM practitioner and "Qi Huang scholar," based on her professional experience of more than 40 years. After more than 20 years of basic and clinical investigation, it has demonstrated its effectiveness in optimizing female reproductive function. We therefore adopt Erzhi Tiangui Fang as a pretreatment for IVF-ET in patients with expected poor ovarian response in order to improve their reproductive outcomes. Outpatient clinics at 10 public tertiary hospitals in the country are involved in the study. It is planned to enroll 480 elderly patients with poor ovarian response between January 2023 and December 2025. The Erzhi Tiangui formula group and placebo group will be randomly assigned in a 1:1 ratio through stratified block randomization. Both groups will use a fixed gonadotrophin releasing hormone (GnRH) antagonist protocol for controlled ovarian hyperstimulation. In IVF cycles, Erzhi tiangui formula and placebo will be administered from day 2 or 3 of the previous menstrual cycle to the trigger day. Approximately 5 to 6 weeks will be required for the intervention to be completed. The primary outcome is the number of retrieved oocytes, i.e., the number of oocytes observed under a microscope after oocyte retrieval monitored by transvaginal ultrasound. Secondary outcomes are the ovarian stimulation outcomes, embryonic laboratory outcomes, pregnancy outcomes, obstetric and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women under 42 years of age with a poor ovarian response (according to the Bologna criteria) .

Exclusion Criteria:

* Individuals with a Body Mass Index (BMI) ≥ 35 Kg/m2.
* Those with a history of unilateral oophorectomy or recurrent pregnancy loss, defined as two or more spontaneous abortions.
* Acceptors of donated oocytes or performed either In vitro Maturation (IVM) or blastocyst biopsy for Preimplantation Genetic Diagnosis (PGD) or Preimplantation Genetic Testing for Aneuploidies (PGT-A).
* Those previously diagnosed with congenital (e.g., mediastinal uterus and double uterus) or acquired (e.g., submucosal myoma and adenomyosis) uterine abnormalities.
* Presence of a non-surgically treated hydrosalpinx or endometrial polyp and an ovarian endometriosis cyst requiring surgery, during ovarian stimulation.
* Allergy to or intolerance of the drugs used in the study.
* Combined contraindications to assisted reproductive technology or pregnancy, such as uncontrolled abnormalities of liver and kidney function, diabetes mellitus (glycosylated haemoglobin ≤7%, fasting blood glucose <10 mmol/L ), hypertension, thyroid disease, symptomatic heart disease, moderate to severe anaemia, history of malignancy or thromboembolism or propensity to thrombosis, severe psychiatric disorder, acute infections of the genitourinary system, sexually transmitted diseases, serious adverse habits such as drug abuse, exposure to teratogenic amounts of radiation, toxins, or drugs (such as prednisone or other hormones, adrenaline, antibiotics, or hypertension, cardiovascular, or antiviral medications) during the active procedure period , and uterine factor infertility or physical illness which prevents the ability to bear a pregnancy.

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of oocyte retrieved | One month
  After oocyte retrieval by transvaginal puncture, the number of collected oocytes was observed microscopically.
Cumulative live birth rate | Eighteen months
  Cumulative live birth rates (CLBR), defined as the proportion of deliveries with at least one live birth per started cycle or per oocyte aspiration, including all fresh and/or frozen embryo transfers until one delivery with a live birth or until all embryos were used.

SECONDARY OUTCOMES:
Cycle cancellation rate | One month
  Cycle cancellation is defined as cycle cancelled before obtaining at least one viable embryo for any reason. And cycle cancellation rate is calculated by dividing the number of women cancelled their cycle before obtaining at least one viable embryo for any reason by the total number of women randomized to the specific group.
Number of Metaphase II (MII) oocytes | One month
  MII oocytes is defined as oocytes retrieved that reach the MII phase.
The number of good quality embryo | One month
  Good quality embryo is defined as embryo that is graded as 6-cell grade 2 (6CII) or better or blastocyst. And good quality embryo rate is calculated by dividing the number of good quality embryo by the total number of embryo obtained after fertilization in the specific group.
Implantation rate | Fourteen months
  Number of gestation sac detected / number of embryo transferred.
Cumulative Clinical pregnancy rate | Fourteen months
  Clinical pregnancy will be diagnosed with the detection of an intrauterine gestation sac. And cumulative clinic pregnancy rate is calculated by the number of women who achieves clinical pregnancy after transfers of all study-specific embryos (within 1 year after randomization) by the total number of women randomized to the specific group.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong, China